CLINICAL TRIAL: NCT06397508
Title: A Randomized, Open-Label, 3-Period, Single-Dose, Cross-Over Study in Healthy Participants to Assess the Relative Bioavailability of AGMB-129 Given as Tablet Formulation Versus the Capsule Reference Formulation and to Assess the Effect of Food on Tablet Formulation
Brief Title: Relative Bioavailability and Effect of Food Study With AGMB-129 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agomab Spain S.L. (Industry)
Responsible Party: Sponsor
Organization: Agomab Therapeutics NV (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: AGMB-129-C103
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1 (Experimental): ABC with A=oral capsule under fed conditions B=oral tablet under fasted conditions C=oral tablet under fed conditions
  Interventions: Drug: AGMB-129
- 2 (Experimental): CAB with A=oral capsule under fed conditions B=oral tablet under fasted conditions C=oral tablet under fed conditions
  Interventions: Drug: AGMB-129
- 3 (Experimental): BCA with A=oral capsule under fed conditions B=oral tablet under fasted conditions C=oral tablet under fed conditions
  Interventions: Drug: AGMB-129
- 4 (Experimental): CBA with A=oral capsule under fed conditions B=oral tablet under fasted conditions C=oral tablet under fed conditions
  Interventions: Drug: AGMB-129
- 5 (Experimental): BAC with A=oral capsule under fed conditions B=oral tablet under fasted conditions C=oral tablet under fed conditions
  Interventions: Drug: AGMB-129
- 6 (Experimental): ACB with A=oral capsule under fed conditions B=oral tablet under fasted conditions C=oral tablet under fed conditions
  Interventions: Drug: AGMB-129

INTERVENTIONS:
Drug: AGMB-129 — Each participant will receive 3 study interventions, 1 in each intervention period

SUMMARY:
This is a single-center, open-label, single-dose, randomized, 3-period cross-over, Phase 1 study in healthy adult participants to assess the BA of AGMB-129 tablet formulation relative to that of the reference capsule formulation and to assess the effect of food on the BA of a single oral dose of the AGMB-129 tablet formulation.

A total of 24 participants will be enrolled. Participants will be randomized to 1 of 6 intervention sequences (Williams design) according to a 6-sequence, 3-period design. In 3 sequential intervention periods, each participant will receive 3 study interventions, 1 in each intervention period. The total duration of involvement for each participant, screening through follow-up, will be approximately 6 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female, between 18 and 55 years old (extremes included) on the date of signing the ICF.
2. Body weight of at least 50.0 kg for men and 45.0 kg for women, and a body mass index (BMI) between 19.0 and 30.0 kg/m2 (extremes included) at screening.
3. Must be in good health based on medical history, physical examination, vital signs, and 12-lead ECG in the opinion of the investigator at screening.
4. Total bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) must be ≤1.5x upper limit of normal (ULN) at screening. Other clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered not clinically significant in the opinion of the investigator. Note: Participants with diagnosed Gilbert's syndrome with total bilirubin >1.5 ULN are eligible for the study if AST and ALT are ≤1.5x ULN.

Key Exclusion Criteria:

1. Known hypersensitivity to AGMB-129 ingredients or history of a significant allergic reaction to AGMB-129 ingredients as determined by the investigator.
2. Positive serology for hepatitis B virus surface antigen (HBsAg) or anti-hepatitis C virus [HCV] antibodies at screening, or history of hepatitis from any cause except for hepatitis A that was resolved at least 3 months prior to the first IP administration.
3. History of or a current immunosuppressive condition, including positive human immunodeficiency virus types 1 or 2 (HIV-1 [2]) antibodies at screening.
4. Current or history of vasculitis, valvular heart disease, or large vessel vascular disease (such as aneurism or dissection) at screening.
5. Any illness, judged by the investigator as clinically significant, in the 3 months prior to the first IP administration.
6. Presence or sequelae of gastrointestinal, liver, kidney (estimated glomerular filtration rate [eGFR] ≤80 mL/min/1.73 m² using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs at screening.
7. History of malignancy within the past 5 years prior to screening, except for excised and curatively treated non-metastatic basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma in situ of cervix which is considered cured with minimal risk of recurrence.
8. History or presence of clinically significant abnormalities detected on 12-lead ECG of either rhythm or conduction, e.g., known long QT syndrome or a QT interval corrected for heart rate according to Fridericia's formula (QTcF) >450 ms detected on the 12-lead ECG at screening or Day 1 predose. A first-degree atrioventricular block will not be considered as a clinically significant abnormality.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Cmax for AGMB-129 | From baseline to Day 3
Cmax for MET-158 | From baseline to Day 3
Cmax for MET-154 | From baseline to Day 3
AUC0-t for AGMB-129 | From baseline to Day 3
AUC0-t for MET-158 | From baseline to Day 3
AUC0-t for MET-154 | From baseline to Day 3
AUC0-∞ for AGMB-447 | From baseline to Day 3
AUC0-∞ for MET-158 | From baseline to Day 3
AUC0-∞ for MET-154 | From baseline to Day 3

SECONDARY OUTCOMES:
Number of participants with adverse events | From Screening to Day 5
  To evaluate the safety and tolerability of AGMB-129 in terms of adverse events at every visit
Number of participants with abnormal clinical laboratory values | From Screening to Day 5
  To evaluate the safety and tolerability of AGMB-129 in terms of abnormal laboratory parameters at every visit
Number of participants with abnormal vital signs | From Screening to Day 5
  To evaluate the safety and tolerability of AGMB-129 in terms of vital signs at every visit
Number of participants with abnormal physical exams | From Screening to Day 5
  To evaluate the safety and tolerability of AGMB-129 in terms of physical exams at every visit

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Wiesel, MD, Study Director — Agomab Therapeutics
Locations (1):
- SGS Belgium, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No